CLINICAL TRIAL: NCT07109063
Title: Psychosocial and Clinical Predictors of Depression, Anxiety, and Stress Among Breast Cancer Patients in Iraq: A Multivariate and Path Modeling Analysis
Brief Title: Psychological Distress in Breast Cancer Patients: A Cross-Sectional Study in Iraq
Status: Completed | Type: Observational
Sponsor: Hameed Adnan Hameed (Other)
Responsible Party: Sponsor-Investigator, Hameed Adnan Hameed, Assistant Lecturer of Clinical Pharmacy / PhD Candidate, Al-Maarif University College
Organization: Al-Maarif University College (Other)
Other Study IDs: BC-Psychology-2025
Record Dates: First submitted 2025-07-29; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Psychological Distress; Depression Anxiety Disorder; Stress (Psychology)
Keywords: Mental Health; Oncology Patients; Cross-Sectional Study; Iraq; Psychosocial Support
MeSH Terms: conditions — Breast Neoplasms; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer Patients Group: This group includes all female patients diagnosed with breast cancer who participated in the cross-sectional survey assessing depression, anxiety, and stress in Anbar, Iraq.

SUMMARY:
This cross-sectional study aims to assess the psychological distress, including depression, anxiety, and stress, among breast cancer patients in Anbar, Iraq. Data were collected using validated questionnaires to evaluate mental health status and associated clinical and demographic factors. The findings will provide insights to improve psychosocial support and patient care in oncology settings

DETAILED DESCRIPTION:
This research is a cross-sectional study conducted to investigate the prevalence and severity of psychological distress, including depression, anxiety, and stress, among breast cancer patients in Anbar, Iraq. The study utilized standardized and validated questionnaires (such as PHQ-9, GAD-7, and Perceived Stress Scale) to assess the mental health status of participants. Data on clinical variables, cancer stage, treatment modalities, and socio-demographic characteristics were collected to identify potential predictors of psychological distress. Statistical analyses were performed to explore associations between psychological outcomes and clinical or demographic factors. The results of this study aim to provide evidence to guide psychosocial interventions and enhance patient care strategies in oncology centers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer
* Female patients aged ≥18 years
* Receiving treatment or follow-up at Anbar Cancer Center
* Willing to provide informed consent

Exclusion Criteria:

* Severe cognitive impairment

  * Inability to complete questionnaires
  * Refusal to participate

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of female breast cancer patients attending Anbar Cancer Center in Iraq for treatment or follow-up during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Depression, Anxiety, and Sleep Disturbances among Breast Cancer Patients | 4 months (January 28, 2025 - May 30, 2025)
  Assessment of psychological distress levels (depression, anxiety, and sleep quality) using PHQ-9, GAD-7, and Pittsburgh Sleep Quality Index questionnaires to evaluate mental health outcomes in breast cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Raghda Roshdy Sayed Hussein, PhD, Clinical pharmacy, Principal Investigator — Faculty of pharmacy, Beni-Suef University
Locations (1):
- Anbar Oncology Center, Ramadi, Al-Anbar Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive patient information and there are no current agreements or resources to enable secure data sharing while ensuring confidentiality

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT07109063/Prot_SAP_000.pdf